CLINICAL TRIAL: NCT01665521
Title: Efficacy Evaluation of the HEART Pathway in Emergency Department Patients With Acute Chest Pain
Acronym: HEART Pathway
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00021074; 12CRP12000001 (Other: American Heart Association)
Record Dates: First submitted 2012-08-07; First posted 2012-08-15 (Estimated); Last update posted 2022-03-04 (Actual); Status verified 2018-08

CONDITIONS: Acute Coronary Syndrome; Chest Pain
Keywords: Acute Coronary Syndrome; Chest pain; Risk Stratification; HEART Pathway; Emergency Department
MeSH Terms: conditions — Acute Coronary Syndrome; Chest Pain; Emergencies

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HEART Pathway (Experimental): The HEART Pathway will be used for real time clinical decision making. Physicians will receive care recommendations according to the HEART Pathway, based on HEART score and serial cardiac biomarkers. This will help physicians identify low-risk patients for early discharge with no objective cardiac testing.
  Interventions: Other: HEART Pathway
- Usual Care (No Intervention): Conventional Care cardiac testing. Patients will undergo cardiac testing as determined by their treating physicians.

INTERVENTIONS:
Other: HEART Pathway — During ED evaluation, patients are randomized to HEART Pathway or usual care arms.
  Arms: HEART Pathway

SUMMARY:
Our research will examine a chest pain care strategy, called the HEART pathway, which is designed to correctly identify Emergency Department patients at high-risk for cardiovascular events, likely to benefit from further testing, and patients at very-low-risk for cardiovascular events, who may be safely discharged home. By using an individual's risk assessment to determining testing, we hope to improve the quality and efficiency of the care delivered to Emergency Department patients with chest pain. Our study will determine if the HEART pathway, which combines a clinical decision rule, the HEART score, and two serial troponin measurements, will reduce stress testing and cardiovascular imaging, decrease hospital length of stay, and reduce cost compared to usual care, while maintaining safety.

DETAILED DESCRIPTION:
Approximately 8-10 million patients complaining of chest pain present to an Emergency Department (ED) annually in the United States. The total cost of chest pain evaluations has been estimated at $5-10 billion annually, yet only 10% of these patients are ultimately diagnosed with an acute coronary syndrome. American College of Cardiology/ American Heart Association (ACC/AHA) guidelines recommend that patients at low-risk for acute coronary syndrome should receive serial cardiac markers followed by objective cardiac testing (stress testing or cardiac imaging). However, many have questioned the value of objective cardiac testing in all low-risk patients.Cardiac testing for all patients at low-risk for acute coronary syndrome (ACS) is not sustainable from a healthcare quality or economic perspective. In addition to increasing costs, objective cardiac testing is associated with a substantial number of false positive and non-diagnostic tests, which lead to additional unnecessary and often invasive procedures.

Implementation of accurate risk stratification care pathways designed to eliminate unnecessary cardiac testing could improve the efficiency and quality of care by decreasing false positive/non-diagnostic testing, radiation, and costs. The HEART pathway, which combines a clinical decision rule, the HEART score, and two serial troponin measurements, is a recently developed care pathway designed to identify chest pain patients for early discharge without objective testing.

Primary Hypothesis: The HEART Pathway, when compared to usual care, will reduce 30 day objective cardiac testing, hospital length of stay, and cost, while maintaining patient safety.

Methods: Participants (n=282) at risk for ACS will be recruited into a clinical trial from Wake Forest Baptist Medical Center (WFBMC) ED. Patients will be equally randomized to HEART Pathway or Usual Care. HEART Pathway participant's treating physician will follow HEART Pathway guidelines for identifying patients to be admitted to the hospital or observation unit for cardiac testing or to be discharged home without testing. Usual Care participant's treating physicians will decide whether the patients should be discharged home or admitted to the hospital or observation unit based on ACC/AHA guidelines without using the HEART pathway.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 21 years
* Chest discomfort or other symptoms consistent with possible ACS
* The treating physician feels the patient could be discharged home if cardiac disease was excluded

Exclusion Criteria:

* New ST-segment elevation in contiguous leads on any electrocardiogram (>/= 1 mV)
* Unstable vitals signs: symptomatic hypotension at the time of enrollment (systolic < 90 mm Hg), tachycardia (HR>120), bradycardia (HR<40), and hypoxemia (<90% pulse-oximetry on room air or normal home oxygen flow rate)
* Terminal diagnosis with life expectancy less than 1 year
* A non-cardiac medical, surgical, or psychiatric illness determined by the provider to require admission, increase risk of objective cardiac testing, or prevent immediate discharge following negative testing.
* Prior enrollment
* Incapacity or unwillingness to provide consent and comply with study procedures
* Non-English speaking

Sub-study I & II

Inclusion Criteria:

* ED attending physicians

Exclusion Criteria:

* ED attending physicians who decline to participate

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2016-02-20 (Actual); Study Completion 2018-01-15 (Actual)

PRIMARY OUTCOMES:
Objective cardiac testing (stress testing or cardiac imaging) within 30 days | 30 Days
  Rate of objective cardiac testing within 30 days

SECONDARY OUTCOMES:
Cost, length of stay, recurrent ED visits and non-index hospitalization for chest pain. | 30 Days
Objective cardiac testing (stress testing or cardiac imaging), cost, length of stay, and recurrent ED visits and non-index hospitalization for chest pain. | 1 Year
Index objective cardiac testing rate | Duration of Index Hospitalization, average of 1 to 2 days
  proportion of patients receiving any stress testing modality, coronary computed tomography angiography, or invasive catheter angiography at the index visit
Index Hospital Admission Rate | Duration of Index Hospitalization, average of 1 to 2 days
  Proportion of patients hospitalized for admission or observation during the index visit
Early discharge rate | Duration of Index Hospitalization, average of 1 to 2 days
  Proportion of patients that are discharged from the Emergency Department without meeting the composite endpoint of index hospital admission or index objective cardiac testing
Composite of 30 day hospital admission and objective cardiac testing | 30 Days

OTHER OUTCOMES:
Major adverse cardiac events (MACE) | 30 Days and 1 Year
Missed MACE | 30 Days and 1 Year
  MACE occurring in patients discharged without objective cardiac testing.
Provider adherence to the HEART Pathway | Duration of Index Hospitalization, average of 1 to 2 days
Inter-rater reliability of the HEART Pathway | Duration of the Index ED visit, less than 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Simon A Mahler, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Wake Forest University Baptist Medical Center - Emergency Department, Winston-Salem, North Carolina, United States

REFERENCES:
- [Background] Rosamond W, Flegal K, Friday G, Furie K, Go A, Greenlund K, Haase N, Ho M, Howard V, Kissela B, Kittner S, Lloyd-Jones D, McDermott M, Meigs J, Moy C, Nichol G, O'Donnell CJ, Roger V, Rumsfeld J, Sorlie P, Steinberger J, Thom T, Wasserthiel-Smoller S, Hong Y; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2007 update: a report from the American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Circulation. 2007 Feb 6;115(5):e69-171. doi: 10.1161/CIRCULATIONAHA.106.179918. Epub 2006 Dec 28. No abstract available. PMID 17194875
- [Background] McCaig LF, Nawar EW. National Hospital Ambulatory Medical Care Survey: 2004 emergency department summary. Adv Data. 2006 Jun 23;(372):1-29. PMID 16841785
- [Background] Owens PL, Barrett ML, Gibson TB, Andrews RM, Weinick RM, Mutter RL. Emergency department care in the United States: a profile of national data sources. Ann Emerg Med. 2010 Aug;56(2):150-65. doi: 10.1016/j.annemergmed.2009.11.022. Epub 2010 Jan 15. PMID 20074834
- [Background] Pope JH, Aufderheide TP, Ruthazer R, Woolard RH, Feldman JA, Beshansky JR, Griffith JL, Selker HP. Missed diagnoses of acute cardiac ischemia in the emergency department. N Engl J Med. 2000 Apr 20;342(16):1163-70. doi: 10.1056/NEJM200004203421603. PMID 10770981
- [Background] Pines JM, Isserman JA, Szyld D, Dean AJ, McCusker CM, Hollander JE. The effect of physician risk tolerance and the presence of an observation unit on decision making for ED patients with chest pain. Am J Emerg Med. 2010 Sep;28(7):771-9. doi: 10.1016/j.ajem.2009.03.019. Epub 2010 Feb 25. PMID 20837253
- [Background] Fleischmann KE, Goldman L, Johnson PA, Krasuski RA, Bohan JS, Hartley LH, Lee TH. Critical pathways for patients with acute chest pain at low risk. J Thromb Thrombolysis. 2002 Apr;13(2):89-96. doi: 10.1023/a:1016246814235. PMID 12101386
- [Background] Roger VL, Go AS, Lloyd-Jones DM, Adams RJ, Berry JD, Brown TM, Carnethon MR, Dai S, de Simone G, Ford ES, Fox CS, Fullerton HJ, Gillespie C, Greenlund KJ, Hailpern SM, Heit JA, Ho PM, Howard VJ, Kissela BM, Kittner SJ, Lackland DT, Lichtman JH, Lisabeth LD, Makuc DM, Marcus GM, Marelli A, Matchar DB, McDermott MM, Meigs JB, Moy CS, Mozaffarian D, Mussolino ME, Nichol G, Paynter NP, Rosamond WD, Sorlie PD, Stafford RS, Turan TN, Turner MB, Wong ND, Wylie-Rosett J; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2011 update: a report from the American Heart Association. Circulation. 2011 Feb 1;123(4):e18-e209. doi: 10.1161/CIR.0b013e3182009701. Epub 2010 Dec 15. PMID 21160056
- [Background] Goldstein JA, Gallagher MJ, O'Neill WW, Ross MA, O'Neil BJ, Raff GL. A randomized controlled trial of multi-slice coronary computed tomography for evaluation of acute chest pain. J Am Coll Cardiol. 2007 Feb 27;49(8):863-71. doi: 10.1016/j.jacc.2006.08.064. Epub 2007 Feb 12. PMID 17320744
- [Background] Farkouh ME, Smars PA, Reeder GS, Zinsmeister AR, Evans RW, Meloy TD, Kopecky SL, Allen M, Allison TG, Gibbons RJ, Gabriel SE. A clinical trial of a chest-pain observation unit for patients with unstable angina. Chest Pain Evaluation in the Emergency Room (CHEER) Investigators. N Engl J Med. 1998 Dec 24;339(26):1882-8. doi: 10.1056/NEJM199812243392603. PMID 9862943
- [Background] Heller GV, Stowers SA, Hendel RC, Herman SD, Daher E, Ahlberg AW, Baron JM, Mendes de Leon CF, Rizzo JA, Wackers FJ. Clinical value of acute rest technetium-99m tetrofosmin tomographic myocardial perfusion imaging in patients with acute chest pain and nondiagnostic electrocardiograms. J Am Coll Cardiol. 1998 Apr;31(5):1011-7. doi: 10.1016/s0735-1097(98)00057-6. PMID 9562001
- [Background] Sprivulis PC, Da Silva JA, Jacobs IG, Frazer AR, Jelinek GA. The association between hospital overcrowding and mortality among patients admitted via Western Australian emergency departments. Med J Aust. 2006 Mar 6;184(5):208-12. doi: 10.5694/j.1326-5377.2006.tb00416.x. PMID 16515429
- [Background] Miro O, Antonio MT, Jimenez S, De Dios A, Sanchez M, Borras A, Milla J. Decreased health care quality associated with emergency department overcrowding. Eur J Emerg Med. 1999 Jun;6(2):105-7. doi: 10.1097/00063110-199906000-00003. PMID 10461551
- [Background] Braunwald E, Antman EM, Beasley JW, Califf RM, Cheitlin MD, Hochman JS, Jones RH, Kereiakes D, Kupersmith J, Levin TN, Pepine CJ, Schaeffer JW, Smith EE 3rd, Steward DE, Theroux P, Gibbons RJ, Alpert JS, Faxon DP, Fuster V, Gregoratos G, Hiratzka LF, Jacobs AK, Smith SC Jr; American College of Cardiology; American Heart Association. Committee on the Management of Patients With Unstable Angina. ACC/AHA 2002 guideline update for the management of patients with unstable angina and non-ST-segment elevation myocardial infarction--summary article: a report of the American College of Cardiology/American Heart Association task force on practice guidelines (Committee on the Management of Patients With Unstable Angina). J Am Coll Cardiol. 2002 Oct 2;40(7):1366-74. doi: 10.1016/s0735-1097(02)02336-7. No abstract available. PMID 12383588
- [Background] Anderson JL, Adams CD, Antman EM, Bridges CR, Califf RM, Casey DE Jr, Chavey WE 2nd, Fesmire FM, Hochman JS, Levin TN, Lincoff AM, Peterson ED, Theroux P, Wenger NK, Wright RS, Smith SC Jr, Jacobs AK, Adams CD, Anderson JL, Antman EM, Halperin JL, Hunt SA, Krumholz HM, Kushner FG, Lytle BW, Nishimura R, Ornato JP, Page RL, Riegel B; American College of Cardiology; American Heart Association Task Force on Practice Guidelines (Writing Committee to Revise the 2002 Guidelines for the Management of Patients With Unstable Angina/Non-ST-Elevation Myocardial Infarction); American College of Emergency Physicians; Society for Cardiovascular Angiography and Interventions; Society of Thoracic Surgeons; American Association of Cardiovascular and Pulmonary Rehabilitation; Society for Academic Emergency Medicine. ACC/AHA 2007 guidelines for the management of patients with unstable angina/non-ST-Elevation myocardial infarction: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (Writing Committee to Revise the 2002 Guidelines for the Management of Patients With Unstable Angina/Non-ST-Elevation Myocardial Infarction) developed in collaboration with the American College of Emergency Physicians, the Society for Cardiovascular Angiography and Interventions, and the Society of Thoracic Surgeons endorsed by the American Association of Cardiovascular and Pulmonary Rehabilitation and the Society for Academic Emergency Medicine. J Am Coll Cardiol. 2007 Aug 14;50(7):e1-e157. doi: 10.1016/j.jacc.2007.02.013. No abstract available. PMID 17692738
- [Background] Ellestad MH, Savitz S, Bergdall D, Teske J. The false positive stress test. Multivariate analysis of 215 subjects with hemodynamic, angiographic and clinical data. Am J Cardiol. 1977 Nov;40(5):681-5. doi: 10.1016/0002-9149(77)90182-5. No abstract available. PMID 920605
- [Background] Bamberg F, Abbara S, Schlett CL, Cury RC, Truong QA, Rogers IS, Nagurney JT, Brady TJ, Hoffmann U. Predictors of image quality of coronary computed tomography in the acute care setting of patients with chest pain. Eur J Radiol. 2010 Apr;74(1):182-8. doi: 10.1016/j.ejrad.2009.03.001. Epub 2009 Apr 5. PMID 19346094
- [Background] Iskandrian AS, Heo J. Appraisal of false positive results in nuclear cardiac imaging. Am Heart J. 1990 Mar;119(3 Pt 1):708-9. doi: 10.1016/s0002-8703(05)80309-6. No abstract available. PMID 2309622
- [Background] Bach DS, Muller DW, Gros BJ, Armstrong WF. False positive dobutamine stress echocardiograms: characterization of clinical, echocardiographic and angiographic findings. J Am Coll Cardiol. 1994 Oct;24(4):928-33. doi: 10.1016/0735-1097(94)90851-6. PMID 7930226
- [Background] Einstein AJ, Henzlova MJ, Rajagopalan S. Estimating risk of cancer associated with radiation exposure from 64-slice computed tomography coronary angiography. JAMA. 2007 Jul 18;298(3):317-23. doi: 10.1001/jama.298.3.317. PMID 17635892
- [Background] Thompson RC, Cullom SJ. Issues regarding radiation dosage of cardiac nuclear and radiography procedures. J Nucl Cardiol. 2006 Jan-Feb;13(1):19-23. doi: 10.1016/j.nuclcard.2005.11.004. No abstract available. PMID 16464713
- [Background] Wagner EH. Chronic disease management: what will it take to improve care for chronic illness? Eff Clin Pract. 1998 Aug-Sep;1(1):2-4. No abstract available. PMID 10345255
- [Background] Six AJ, Backus BE, Kelder JC. Chest pain in the emergency room: value of the HEART score. Neth Heart J. 2008 Jun;16(6):191-6. doi: 10.1007/BF03086144. PMID 18665203
- [Background] Backus BE, Six AJ, Kelder JC, Mast TP, van den Akker F, Mast EG, Monnink SH, van Tooren RM, Doevendans PA. Chest pain in the emergency room: a multicenter validation of the HEART Score. Crit Pathw Cardiol. 2010 Sep;9(3):164-9. doi: 10.1097/HPC.0b013e3181ec36d8. PMID 20802272
- [Background] Mahler SA, Hiestand BC, Goff DC Jr, Hoekstra JW, Miller CD. Can the HEART score safely reduce stress testing and cardiac imaging in patients at low risk for major adverse cardiac events? Crit Pathw Cardiol. 2011 Sep;10(3):128-33. doi: 10.1097/HPC.0b013e3182315a85. PMID 21989033
- [Background] Than M, Cullen L, Reid CM, Lim SH, Aldous S, Ardagh MW, Peacock WF, Parsonage WA, Ho HF, Ko HF, Kasliwal RR, Bansal M, Soerianata S, Hu D, Ding R, Hua Q, Seok-Min K, Sritara P, Sae-Lee R, Chiu TF, Tsai KC, Chu FY, Chen WK, Chang WH, Flaws DF, George PM, Richards AM. A 2-h diagnostic protocol to assess patients with chest pain symptoms in the Asia-Pacific region (ASPECT): a prospective observational validation study. Lancet. 2011 Mar 26;377(9771):1077-84. doi: 10.1016/S0140-6736(11)60310-3. PMID 21435709
- [Background] Than M, Cullen L, Aldous S, Parsonage WA, Reid CM, Greenslade J, Flaws D, Hammett CJ, Beam DM, Ardagh MW, Troughton R, Brown AF, George P, Florkowski CM, Kline JA, Peacock WF, Maisel AS, Lim SH, Lamanna A, Richards AM. 2-Hour accelerated diagnostic protocol to assess patients with chest pain symptoms using contemporary troponins as the only biomarker: the ADAPT trial. J Am Coll Cardiol. 2012 Jun 5;59(23):2091-8. doi: 10.1016/j.jacc.2012.02.035. Epub 2012 May 9. PMID 22578923
- [Background] Backus BE, Six AJ, Kelder JC, Bosschaert MA, Mast EG, Mosterd A, Veldkamp RF, Wardeh AJ, Tio R, Braam R, Monnink SH, van Tooren R, Mast TP, van den Akker F, Cramer MJ, Poldervaart JM, Hoes AW, Doevendans PA. A prospective validation of the HEART score for chest pain patients at the emergency department. Int J Cardiol. 2013 Oct 3;168(3):2153-8. doi: 10.1016/j.ijcard.2013.01.255. Epub 2013 Mar 7. PMID 23465250
- [Background] Hollander JE. Risk stratification of emergency department patients with chest pain: the need for standardized reporting guidelines. Ann Emerg Med. 2004 Jan;43(1):68-70. doi: 10.1016/s0196-0644(03)00726-1. No abstract available. PMID 14707943
- [Background] Peacock WF, Nagurney J, Birkhahn R, Singer A, Shapiro N, Hollander J, Glynn T, Nowak R, Safdar B, Miller C, Peberdy M, Counselman F, Chandra A, Kosowsky J, Neuenschwander J, Schrock J, Plantholt S, Lewandrowski E, Wong V, Kupfer K, Diercks D. Myeloperoxidase in the diagnosis of acute coronary syndromes: the importance of spectrum. Am Heart J. 2011 Nov;162(5):893-9. doi: 10.1016/j.ahj.2011.08.017. PMID 22093206
- [Background] Hess EP, Brison RJ, Perry JJ, Calder LA, Thiruganasambandamoorthy V, Agarwal D, Sadosty AT, Silvilotti ML, Jaffe AS, Montori VM, Wells GA, Stiell IG. Development of a clinical prediction rule for 30-day cardiac events in emergency department patients with chest pain and possible acute coronary syndrome. Ann Emerg Med. 2012 Feb;59(2):115-25.e1. doi: 10.1016/j.annemergmed.2011.07.026. Epub 2011 Sep 1. PMID 21885156
- [Background] Kirby SE, Dennis SM, Jayasinghe UW, Harris MF. Patient related factors in frequent readmissions: the influence of condition, access to services and patient choice. BMC Health Serv Res. 2010 Jul 21;10:216. doi: 10.1186/1472-6963-10-216. PMID 20663141
- [Background] Herlitz J, Karlson BW, Sjolin M. Re-admissions among patients with acute chest pain who were discharged from the emergency department. Eur J Emerg Med. 1996 Mar;3(1):31-5. doi: 10.1097/00063110-199603000-00006. PMID 8886668
- [Background] Herlitz J, Karlson BW, Lindqvist J, Sjolin M. Characteristics and long-term outcome of patients with acute chest pain or other symptoms raising suspicion of acute myocardial infarction in relation to whether they were hospitalized or directly discharged from the emergency department. Coron Artery Dis. 2002 Feb;13(1):37-43. doi: 10.1097/00019501-200202000-00005. PMID 11917197
- [Background] Meyer MC, Mooney RP, Sekera AK. A critical pathway for patients with acute chest pain and low risk for short-term adverse cardiac events: role of outpatient stress testing. Ann Emerg Med. 2006 May;47(5):427-35. doi: 10.1016/j.annemergmed.2005.10.010. Epub 2006 Feb 8. PMID 16631982
- [Background] Richards D, Meshkat N, Chu J, Eva K, Worster A. Emergency department patient compliance with follow-up for outpatient exercise stress testing: a randomized controlled trial. CJEM. 2007 Nov;9(6):435-40. doi: 10.1017/s1481803500015463. PMID 18072989
- [Background] Cannon CP, Hoekstra JW, Larson DM, Carter RD, Cornish J, Karcher RB, Mencia WA, Berry CA, Stowell SA. Physician practice patterns in acute coronary syndromes: an initial report of an individual quality improvement program. Crit Pathw Cardiol. 2010 Mar;9(1):23-9. doi: 10.1097/HPC.0b013e3181d09d2d. PMID 20215907
- [Background] Blomkalns AL, Roe MT, Peterson ED, Ohman EM, Fraulo ES, Gibler WB. Guideline implementation research: exploring the gap between evidence and practice in the CRUSADE Quality Improvement Initiative. Acad Emerg Med. 2007 Nov;14(11):949-54. doi: 10.1197/j.aem.2007.06.017. PMID 17967956
- [Background] Miller CD, Hoekstra JW, Lefebvre C, Blumstein H, Hamilton CA, Harper EN, Mahler S, Diercks DB, Neiberg R, Hundley WG. Provider-directed imaging stress testing reduces health care expenditures in lower-risk chest pain patients presenting to the emergency department. Circ Cardiovasc Imaging. 2012 Jan;5(1):111-8. doi: 10.1161/CIRCIMAGING.111.965293. Epub 2011 Nov 29. PMID 22128195
- [Background] Mahler S, Nwanaji-Enwerem J, Miller C, Hoekstra J, Goff D. Coronary Computed Tomography Angiography Decreases Length of Stay in Patients With Acute Chest Pain Compared to Stress Testing: Does Time of Patient Presentation Affect This Relationship? J Am Coll Cardiol 2011;57:E666.
- [Background] Hollander JE, Blomkalns AL, Brogan GX, Diercks DB, Field JM, Garvey JL, Gibler WB, Henry TD, Hoekstra JW, Holroyd BR, Hong Y, Kirk JD, O'Neil BJ, Jackson RE; Multidisciplinary Standardized Reporting Criteria Task Force. Standardized reporting guidelines for studies evaluating risk stratification of ED patients with potential acute coronary syndromes. Acad Emerg Med. 2004 Dec;11(12):1331-40. doi: 10.1197/j.aem.2004.08.033. No abstract available. PMID 15576525
- [Background] Adams G, Abusaid G, Lee B, Maynard C, Campbell P, Wagner G, Barbagelata A. From theory to practice: implementation of pre-hospital electrocardiogram transmission in ST-elevation myocardial infarction - a multicenter experience. J Invasive Cardiol. 2010 Nov;22(11):520-5. PMID 21041847
- [Background] Abcarian PW, Sweet JD, Watabe JT, Yoon HC. Role of a quantitative D-dimer assay in determining the need for CT angiography of acute pulmonary embolism. AJR Am J Roentgenol. 2004 Jun;182(6):1377-81. doi: 10.2214/ajr.182.6.1821377. PMID 15149977
- [Background] Corwin MT, Donohoo JH, Partridge R, Egglin TK, Mayo-Smith WW. Do emergency physicians use serum D-dimer effectively to determine the need for CT when evaluating patients for pulmonary embolism? Review of 5,344 consecutive patients. AJR Am J Roentgenol. 2009 May;192(5):1319-23. doi: 10.2214/AJR.08.1346. PMID 19380556
- [Background] Yin F, Wilson T, Della Fave A, Larsen M, Yoon J, Nugusie B, Freeland H, Chow RD. Inappropriate use of D-dimer assay and pulmonary CT angiography in the evaluation of suspected acute pulmonary embolism. Am J Med Qual. 2012 Jan-Feb;27(1):74-9. doi: 10.1177/1062860611407907. Epub 2011 Jun 10. PMID 21666066
- [Background] Anderson JL, Adams CD, Antman EM, Bridges CR, Califf RM, Casey DE Jr, Chavey WE 2nd, Fesmire FM, Hochman JS, Levin TN, Lincoff AM, Peterson ED, Theroux P, Wenger NK, Wright RS, Jneid H, Ettinger SM, Ganiats TG, Lincoff AM, Philippides GJ, Zidar JP; American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. 2012 ACCF/AHA focused update incorporated into the ACCF/AHA 2007 guidelines for the management of patients with unstable angina/non-ST-elevation myocardial infarction: a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. Circulation. 2013 Jun 11;127(23):e663-828. doi: 10.1161/CIR.0b013e31828478ac. Epub 2013 Apr 29. No abstract available. PMID 23630129
- [Background] Wright RS, Anderson JL, Adams CD, Bridges CR, Casey DE Jr, Ettinger SM, Fesmire FM, Ganiats TG, Jneid H, Lincoff AM, Peterson ED, Philippides GJ, Theroux P, Wenger NK, Zidar JP, Jacobs AK. 2011 ACCF/AHA Focused Update of the Guidelines for the Management of Patients With Unstable Angina/ Non-ST-Elevation Myocardial Infarction (Updating the 2007 Guideline): a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. Circulation. 2011 May 10;123(18):2022-60. doi: 10.1161/CIR.0b013e31820f2f3e. Epub 2011 Mar 28. No abstract available. PMID 21444889
- [Background] O'Connor RE, Bossaert L, Arntz HR, Brooks SC, Diercks D, Feitosa-Filho G, Nolan JP, Vanden Hoek TL, Walters DL, Wong A, Welsford M, Woolfrey K; Acute Coronary Syndrome Chapter Collaborators. Part 9: Acute coronary syndromes: 2010 International Consensus on Cardiopulmonary Resuscitation and Emergency Cardiovascular Care Science With Treatment Recommendations. Circulation. 2010 Oct 19;122(16 Suppl 2):S422-65. doi: 10.1161/CIRCULATIONAHA.110.985549. No abstract available. PMID 20956257
- [Background] Miller CD, Hwang W, Case D, Hoekstra JW, Lefebvre C, Blumstein H, Hamilton CA, Harper EN, Hundley WG. Stress CMR imaging observation unit in the emergency department reduces 1-year medical care costs in patients with acute chest pain: a randomized study for comparison with inpatient care. JACC Cardiovasc Imaging. 2011 Aug;4(8):862-70. doi: 10.1016/j.jcmg.2011.04.016. PMID 21835378
- [Background] Kline JA, Mitchell AM, Runyon MS, Jones AE, Webb WB. Electronic medical record review as a surrogate to telephone follow-up to establish outcome for diagnostic research studies in the emergency department. Acad Emerg Med. 2005 Nov;12(11):1127-33. doi: 10.1197/j.aem.2005.04.012. Epub 2005 Sep 15. PMID 16166598
- [Background] Miller CD, Hwang W, Hoekstra JW, Case D, Lefebvre C, Blumstein H, Hiestand B, Diercks DB, Hamilton CA, Harper EN, Hundley WG. Stress cardiac magnetic resonance imaging with observation unit care reduces cost for patients with emergent chest pain: a randomized trial. Ann Emerg Med. 2010 Sep;56(3):209-219.e2. doi: 10.1016/j.annemergmed.2010.04.009. Epub 2010 May 31. PMID 20554078
- [Background] Thygesen K, Alpert JS, White HD; Joint ESC/ACCF/AHA/WHF Task Force for the Redefinition of Myocardial Infarction; Jaffe AS, Apple FS, Galvani M, Katus HA, Newby LK, Ravkilde J, Chaitman B, Clemmensen PM, Dellborg M, Hod H, Porela P, Underwood R, Bax JJ, Beller GA, Bonow R, Van der Wall EE, Bassand JP, Wijns W, Ferguson TB, Steg PG, Uretsky BF, Williams DO, Armstrong PW, Antman EM, Fox KA, Hamm CW, Ohman EM, Simoons ML, Poole-Wilson PA, Gurfinkel EP, Lopez-Sendon JL, Pais P, Mendis S, Zhu JR, Wallentin LC, Fernandez-Aviles F, Fox KM, Parkhomenko AN, Priori SG, Tendera M, Voipio-Pulkki LM, Vahanian A, Camm AJ, De Caterina R, Dean V, Dickstein K, Filippatos G, Funck-Brentano C, Hellemans I, Kristensen SD, McGregor K, Sechtem U, Silber S, Tendera M, Widimsky P, Zamorano JL, Morais J, Brener S, Harrington R, Morrow D, Lim M, Martinez-Rios MA, Steinhubl S, Levine GN, Gibler WB, Goff D, Tubaro M, Dudek D, Al-Attar N. Universal definition of myocardial infarction. Circulation. 2007 Nov 27;116(22):2634-53. doi: 10.1161/CIRCULATIONAHA.107.187397. Epub 2007 Oct 19. No abstract available. PMID 17951284
- [Background] Myocardial infarction redefined--a consensus document of The Joint European Society of Cardiology/American College of Cardiology Committee for the redefinition of myocardial infarction. Eur Heart J. 2000 Sep;21(18):1502-13. doi: 10.1053/euhj.2000.2305. PMID 10973764
- [Background] Geleijnse ML, Fioretti PM, Roelandt JR. Methodology, feasibility, safety and diagnostic accuracy of dobutamine stress echocardiography. J Am Coll Cardiol. 1997 Sep;30(3):595-606. doi: 10.1016/s0735-1097(97)00206-4. PMID 9283514
- [Background] Christenson J, Innes G, McKnight D, Boychuk B, Grafstein E, Thompson CR, Rosenberg F, Anis AH, Gin K, Tilley J, Wong H, Singer J. Safety and efficiency of emergency department assessment of chest discomfort. CMAJ. 2004 Jun 8;170(12):1803-7. doi: 10.1503/cmaj.1031315. PMID 15184334
- [Background] Gomez MA, Anderson JL, Karagounis LA, Muhlestein JB, Mooers FB. An emergency department-based protocol for rapidly ruling out myocardial ischemia reduces hospital time and expense: results of a randomized study (ROMIO). J Am Coll Cardiol. 1996 Jul;28(1):25-33. doi: 10.1016/0735-1097(96)00093-9. PMID 8752791
- [Derived] Mahler SA, Riley RF, Hiestand BC, Russell GB, Hoekstra JW, Lefebvre CW, Nicks BA, Cline DM, Askew KL, Elliott SB, Herrington DM, Burke GL, Miller CD. The HEART Pathway randomized trial: identifying emergency department patients with acute chest pain for early discharge. Circ Cardiovasc Qual Outcomes. 2015 Mar;8(2):195-203. doi: 10.1161/CIRCOUTCOMES.114.001384. Epub 2015 Mar 3. PMID 25737484
- See also: Wake Forest Baptist Health — http://www.wakehealth.edu